CLINICAL TRIAL: NCT01306500
Title: Effect of Gastric Lavage in Preventing Feeding Problems in Late Preterm and Term Neonates Born With Meconium Stained Amniotic Fluid : A Randomized Controlled Trial
Brief Title: Effect of Gastric Lavage in Preventing Feeding Problems in Babies Born With Meconium Stained Amniotic Fluid
Acronym: GLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr Sushma Nangia, Professor of Pediatrics, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LHMC/035/2010/GLAM
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Gastritis of Newborn; Other Vomiting of Newborn; Meconium in Amniotic Fluid
Keywords: Gastric lavage; Neonate; Meconium stained amniotic fluid; Feeding problems
MeSH Terms: interventions — Gastric Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastric lavage Group (Experimental): In neonates randomized to intervention Group (gastric lavage group) gastric lavage was done in the labor room after initial stabilization
  Interventions: Procedure: Gastric lavage
- No gastric lavage (No Intervention): Neonates randomized to 'No gastric lavage group' will receive supportive treatment as per standard unit protocol.

INTERVENTIONS:
Procedure: Gastric lavage — 8 Fr feeding tube was inserted orally with length equal to distance from the bridge of the nose to the earlobe and from the earlobe to a point halfway between the xiphoid process and the umbilicus. 20ml normal saline was used for gastric lavage. It was ensured that entire amount of normal saline used was removed from stomach.
  Arms: Gastric lavage Group

SUMMARY:
The purpose of the study is to evaluate the role of gastric lavage in preventing feeding problems in babies born through meconium stained amniotic fluid. It is a routine practice in many hospitals to perform gastric lavage in all babies born with meconium stained amniotic fluid after stabilisation without any supporting evidence. It is believed that meconium is an irritant and its presence in stomach causes gastritis and vomiting and hence the basis for this practice. Orogastric tube insertion and subsequent gastric lavage is not without complications. Potential complications will be prevented and health resources will be saved if this procedure is not proven to be beneficial. Therefore the investigators decided to study if gastric lavage reduces incidence of vomiting and other feeding difficulties as well as incidence of respiratory difficulties in babies born with MSAF.

DETAILED DESCRIPTION:
Meconium passage in newborn infants is a developmentally programmed event normally occurring within first 24-48 hours of birth. The meconium staining of amniotic fluid occurs in 12% of all live births per annuum.

The routine use of gastric lavage in MSAF babies has been advocated for a long time as a part of the conventional treatment. Meconium in stomach is hypothesized to act as an irritant and cause vomiting and retching. Surprisingly this recommendation is also made in some textbooks without supporting evidence.

Orogastric tube insertion and subsequent gastric lavage can cause complications like bradycardia, apnea, vomiting, trauma, aspiration and esophageal or gastric perforations. Some researchers have found that gastric suction done at birth is associated with long term risk for functional intestinal disorder. The sequence of prefeeding behaviour is disrupted in children who undergo gastric suction and it can delay initiation of breast feeding. Small elevation in mean arterial blood pressure, increased retching have also been reported The role of gastric lavage in preventing feeding problems and secondary meconium aspiration syndrome has not been systematically evaluated. If this procedure is not proven to be beneficial it will prevent potential complications which may arise due to it in a significant number of babies. Also in a resource limited country the cost of materials required and time of medical personnel will be saved. Hence the purpose of this prospective randomized controlled trial is to compare the incidence of feeding problems and secondary meconium aspiration syndrome, in gastric lavage group vs no lavage group.

ELIGIBILITY:
Inclusion Criteria:

* Gestation > 34 weeks
* Meconium staining of amniotic fluid
* Vigorous babies

Exclusion Criteria:

* Major Congenital malformation
* Non vigorous babies
* Refusal of consent

Ages: 2 Minutes to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 538 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Feeding problems | Till discharge from hospital
  Feeding problems were considered to be present
  1. Mother or caretaker gave history of retching, vomiting or both.
  2. Nursing staff or resident on duty observed vomiting, retching or both

SECONDARY OUTCOMES:
Secondary meconium aspiration syndrome | Till discharge from hospital
  Presence of tachypnea or respiratory distress in a previously well baby following vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Principal Investigator — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India